CLINICAL TRIAL: NCT06722586
Title: Sirolimus Monotherapy in the Treatment of Antiphospholipid Antibody Related Thrombocytopenia: a Multicenter Randomized, Double Blind, Placebo Controlled, Clinical Trial
Brief Title: Sirolimus Monotherapy in the Treatment of Antiphospholipid Antibody Related Thrombocytopenia
Acronym: SMART
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: North China Pharmaceutical Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Zhuoli ZHANG, MD, PhD, Director of Rheumatology and Immunology Department, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMART_V2.2
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-01

CONDITIONS: Antiphospholipid (aPL)-Positive; Thrombocytopaenia
Keywords: antiphospholipid; thrombocytopaenia; sirolimus; rapamycin
MeSH Terms: conditions — Thrombocytopenia | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Sirolimus two pills (1mg) per day
  Interventions: Drug: Sirolimus
- Control (Placebo Comparator): Placebo two pills per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — Sirolimus two pills (1mg) per day
  Other Names: Rapamycin; mTOR inhibitor
  Arms: Treatment
Drug: Placebo — Placebo two pills per day
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn the efficacy and safety of sirolimus in the treatment of anti-phospholipid antibody associated thrombocytopenia. The patients would be followed at 2 weeks, 1 month, 3 months, and 6 months after the enrollment. The main questions it aims to answer are the differences between sirolimus and control group at below outcomes:

Primary outcome: the overall response rate at 6 months Secondary outcome: the complete response rate at 6 months the partial response rate at 6 months the change of anti-phospholipid antibody titers the change of oral glucocorticoids dosage Other pre-defined outcome: the dropout rate within 6 months Participants will receive either sirolimus 1mg per day or placebo.

DETAILED DESCRIPTION:
Complete response: the platelet count is more that 100×10^9/L Partial response: If the platelet count is less than 100×10^9/L, it should be more than 2 times of the baseline count Overall response: both complete and partial response

ELIGIBILITY:
Inclusion Criteria:

* persistent positive of antiphospholipid antibody (either lupus anticoagulant, anti-cardiolipin antibody, or anti-b2GP1 antibody, at least two times with 12 weeks apart)
* persistent thrombocytopenia (30-100×10^9/L, at least for 2 weeks)

Eligible concomitant treatment:

* prednisone or equivalent dose less than 10mg per day is allowed, and dose should be stable for more than 2 weeks
* hydroxychloroquine less than 400mg per day is allowed, and dose should be stable for more than 1 month
* anti-platelet and/or anti-coagulant therapy is allowed, and strength should be the stable for 1 week
* these following therapies should be discontinued for more than 5 half-lives before the enrollment, including thrombopoietin or thrombopoietin receptor antagonist, intravenous immunoglobulin, immunosuppressants, B cell inhibitors (Belimumab or Talitacicept) and B cell depletion therapy (Rituximab or Obinutuzumab).

Exclusion Criteria:

* fulling the criteria of other connective tissue disease other than antiphospholipid syndrome
* received oral/intravenous antibiotics within 2 weeks before the enrollment.
* new onset of thrombosis within 4 weeks before the enrollment.
* apparent bleeding tendency.
* life or organ threatening manifestations, includes but not limit to catastrophic antiphospholipid syndrome and thrombotic microangiopathy.
* liver and renal dysfunction: ALT or AST more than three times of upper limit of normal range; eGFR<40mL/min/1.73m^2
* hematocytopenia: WBC<3.0×10^9/L, Hb<100g/L.
* uncontrollable hyperlipidemia: low density lipoprotein cholesterol>3.1 mmol/L, triglycerides>2.3 mmol/L after lipid lowering therapy.
* current active infection
* women in pregnancy and postpartum period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall response | From enrollment to the end of treatment at 6 months
  Both complete response and partial response

SECONDARY OUTCOMES:
Complete response | From enrollment to the end of treatment at 6 months
  Platelet count more than 100×10^9/L
Partial response | From enrollment to the end of treatment at 6 months
  If the platelet count is less than 100×10^9/L, it should be more than 2 times of the baseline platelet count
The change of antiphospholipid antibodies titers | From enrollment to the end of treatment at 6 months
  The changes of titers of antiphospholipid antibodies comparing to that of baseline
The change of oral glucocorticoids dosage | From enrollment to the end of treatment at 6 months
  The differences of oral glucocorticoids dosage change between two groups

OTHER OUTCOMES:
Dropout rate | From enrollment to the end of treatment at 6 months
  The differences of dropout rates between two groups

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Qilu Hospital of Shandong University, Jinan, Shangdong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The 1st Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Chao-Yang Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Shijitan Hospital, Beijing
  - Shanghai Renji Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided